CLINICAL TRIAL: NCT01525446
Title: Proton Stereotactic Body Radiation Therapy (SBRT) for Medically Inoperable, Peripheral Early-Stage Non-Small Cell Lung Cancer (NSCLC): A Pilot Study
Brief Title: Proton Stereotactic Body Radiation Therapy for Early-Stage Non-Small Cell Lung Cancer
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Henning Willers, M.D., Attending Radiation Oncologist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-021
Record Dates: First submitted 2011-07-19; First posted 2012-02-03 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SBRT with proton beam radiation (Experimental): 4 consecutive days for the delivery of 48 Gy (tumors 3 cm or less) or 5 consecutive days for the delivery of 60 Gy (tumors of > 3 cm)
  Interventions: Radiation: SBRT with proton beam radiation

INTERVENTIONS:
Radiation: SBRT with proton beam radiation — 4 consecutive days for the delivery of 48 Gy (tumors 3 cm or less) or 5 consecutive days for the delivery of 60 Gy (tumors of > 3 cm)

SUMMARY:
Stereotactic body radiation therapy (SBRT) is a special form of treatment which pinpoints high doses of radiation directly to cancer. Standard radiation (or photon radiation) is commonly used for SBRT to treat Non-Small Cell Lung Cancer (NSCLC). Proton beam radiation is a special type of radiation only available at a few institutions in the US and has not been previously used in SBRT to treat NSCLC. The use of protons for SBRT may improve the accuracy of the treatment and may help to minimize the dose delivered unnecessarily to healthy tissue.

In this study, the investigators are evaluating the safety and effectiveness of proton-based SBRT for early-stage NSCLC located in the periphery of the lung.

DETAILED DESCRIPTION:
Subjects will undergo an electronic navigational bronchoscopy (ENB) during which three markers will be placed around their tumor which will guide the delivery of proton beam radiation to their with more precision and accuracy.

Subjects will receive a CT scan to obtain images to plan radiation treatment. Proton radiation will be delivered daily (4 or 5 consecutive days) on an outpatient basis at Massachusetts General Hospital.

After the final dose of proton radiation subjects will be followed for 5 years. Subjects will be asked to return at 3 months, and then every 3 months until 2 years, and then every 6 months until 5 years. Subjects will receive a chest CT, tumor assessment by CT or PET, chest x-ray, pulmonary function tests and a physical exam.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (need not be newly diagnosed)
* Stage clinical T1 N0 M0 or T2 N0 M0
* NSCLC must be limited to a single lesion
* NSCLC must be peripherally located (> 2 cm from proximal bronchial tree and > 1 cm from mediastinal pleura)
* NSCLC must be considered medically inoperable
* Life expectancy greater than 6 months

Exclusion Criteria:

* Pregnant or breastfeeding
* Prior radiation therapy to the lungs or mediastinum
* Prior malignancy in the last 2 years unless treated definitively and disease free or carcinoma in situ or early stage skin cancers that have been definitively treated
* Receiving other study agents or other types of cancer therapy
* Uncontrolled intercurrent illness
* Pacemaker or defibrillator-dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety | 2 years
  To establish the feasibility and safety of fiducials placement by electromagnetic navigational bronchoscopy (ENB)
Safety and tolerability | 2 years
  Frequency of radiation pneumonitis in participants treated with proton radiation

SECONDARY OUTCOMES:
Toxicity | 2 years
  Describe the acute and late toxicities of treatment using CTCAE v4.0
Efficacy | 2 years
  To describe radiological tumor responses
Disease Free survival | 2 years
  To calculate local, regional, and distant failure rates
Overall survival | 2 years
  To calculate the overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Henning Willers, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States